CLINICAL TRIAL: NCT00654927
Title: Phase 3 Open-Label Extension Study to Evaluate the Safety, Tolerability and Activity of Oral Fampridine-SR in Patients With Multiple Sclerosis
Brief Title: Open-Label Extension Study to Evaluate the Safety, Tolerability and Activity of Oral Fampridine-SR in Patients With Multiple Sclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Acorda Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS-F202 EXT
Record Dates: First submitted 2008-04-04; First posted 2008-04-09 (Estimated); Results first posted 2012-02-29 (Estimated); Last update posted 2012-03-02 (Estimated); Status verified 2012-01

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; MS; walking; leg strength; demyelination
MeSH Terms: conditions — Multiple Sclerosis; Demyelinating Diseases | interventions — 4-Aminopyridine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Fampridine-SR b.i.d. (Twice Daily) — Dosage form - tablets.
  Other Names: 4-aminopyridine

SUMMARY:
The purpose of this study is to evaluate the long-term safety, tolerability and activity of Fampridine-SR in subjects with multiple sclerosis who have previously participated in either an Acorda Therapeutics or an Elan Corporation sponsored protocol. Subjects are eligible regardless of whether they received active drug or placebo during their participation in the previous study.

DETAILED DESCRIPTION:
Under the original protocol, patients were to have their treatment dose titrated upwards from a starting dose of 10mg b.i.d. to 15mg b.i.d. and then to a stable (maintenance) dose of 20mg b.i.d. The protocol was subsequently revised to lower the maximum maintenance dose. In the most current protocol, all patients were down-titrated to 10mg b.i.d. and maintained at this dose for the greater part of the duration of the study.

Multiple Sclerosis (MS) is a disorder of the body's immune system that affects the central nervous system (CNS). Normally, nerve fibers carry electrical impulses through the spinal cord, providing communication between the brain and the arms and legs. In people with MS, the fatty sheath that surrounds and insulates the nerve fibers (called "myelin") deteriorates, causing nerve impulses to be slowed or stopped. As a result, patients with MS may experience periods of muscle weakness and other symptoms such as numbness, loss of vision, loss of coordination, paralysis, spasticity, mental and physical fatigue and a decrease in the ability to think and/or remember. These periods of illness may come (exacerbations) and go (remissions). Fampridine-SR is an experimental drug that has been reported to possibly improve muscle strength and walking ability for some people with MS. This study will evaluate the effects and possible risks of taking Fampridine-SR in MS patients over a long period of time.

ELIGIBILITY:
Inclusion Criteria:

* The subject must have been previously enrolled in an Acorda Therapeutics or an Elan Corporation sponsored study for multiple sclerosis and received either Fampridine or placebo.
* The subject must have multiple sclerosis as determined by the Principal Investigator.
* The subject, male or female, must be at least 18 years of age. Any subject who is now over the age of 70 must be in good overall health in the judgment of the Investigator.
* The subject must be of adequate cognitive function, as judged by the Investigator.
* Any subject who is female and of childbearing potential, regardless of sexual activity, must have a negative urine pregnancy test at the Screening Visit.

Exclusion Criteria:

* The subject is a female who is either pregnant or breastfeeding, or of child-bearing potential, who, if engaged in active heterosexual relations and has not had a hysterectomy or bilateral oophorectomy, would not use one of the following birth control methods: tubal ligation, implantable contraception device, oral, injectable or transdermal contraceptive, barrier method or sexual activity restricted to vasectomized partner.
* The subject withdrew from a previous Fampridine study because of a Serious Adverse Event that was possibly, probably or definitely related to Fampridine.
* The subject has a history of seizures or has evidence of past, or possible, epileptiform activity on an EEG.
* The subject has either a clinically significant abnormal ECG or laboratory value(s) at the Screening Visit, as judged by the Investigator
* The subject has angina, uncontrolled hypertension, clinically significant cardiac arrhythmias, or any other clinically significant cardiovascular abnormality, as judged by the Investigator.
* The subject has a known allergy to pyridine-containing substances or any of the inactive ingredients of the Fampridine tablet
* The subject has received an investigational drug, except for Fampridine- SR (or matching placebo) under Protocol MS-F202, within 30 days prior to the Screening Visit; or the subject is scheduled to enroll in an investigational drug trial at any time during this study.
* The subject has received compounded 4-aminopyridine (4-AP) within 14 days of the Screening Visit.
* The subject has had an onset of an MS exacerbation within 30 days prior to the Screening Visit, or, if in the judgment of the Investigator, has not stabilized from a prior exacerbation episode.
* The subject has started on a concomitant medication regimen for an underlying disease/symptom within the past 7 days; or has started an interferon or chemotherapeutic agent for multiple sclerosis within the past 4 weeks.
* The subject has a history of drug or alcohol abuse within the past year.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2003-11; Primary Completion 2011-01 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Faust, Study Director — Acorda Therapeutics
Locations (22):
- United States (20):
  - Barrow Neurology Clinic, St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - USC, Keck School of Medicine Health Care Consultation Center, Los Angeles, California
  - Shepherd Center, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Maryland Center for MS, Baltimore, Maryland
  - The Schapiro Center for MS, Golden Valley, Minnesota
  - Washington University School of Medicine, Div. of Rehab/Neurology, St Louis, Missouri
  - Gimbel MS Center at Holy Name Hospital, Teaneck, New Jersey
  - University of Mexico, MIND Imaging Center, Albuquerque, New Mexico
  - Maimonides MS Care Center, Brooklyn, New York
  - Corinne Goldsmith Dickinson Center for MS, New York, New York
  - University of Rochester, Rochester, New York
  - SUNY Stony Brook, Stony Brook, New York
  - CMC - Neuroscience & Spine Institute, Division of Neurology, Charlotte, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University MS Center, Columbus, Ohio
  - Oregon Health & Science University, MS Center of Oregon, UHS-42, Portland, Oregon
  - Thomas Jefferson University Physicians, Philadelphia, Pennsylvania
  - University of Texas-Houston, Houston, Texas
  - MS Center at Evergreen, Kirkland, Washington
- Canada (2):
  - Foothills Medical Center, Calgary, Alberta
  - St. Michael's Hospital, Toronto, Ontario

REFERENCES:
- See also: (Click here for more information about Fampridine-SR clinical trials) — http://www.acorda.com/clinical.asp

RESULTS

PARTICIPANT FLOW:
Groups:
- Fampridine-SR b.i.d. (Twice Daily): All subjects (N=177) received 10mg b.i.d. Tablets.
  (N=175) subjects received 15mg b.i.d and (N=7) subjects received 20mg b.i.d at some point in the study.
Period: Overall Study
Arm/Group | Fampridine-SR b.i.d. (Twice Daily)
Started | 177
Completed | 70
Not Completed | 107

BASELINE CHARACTERISTICS:
Arm/Group | Fampridine-SR b.i.d. (Twice Daily)
Number analyzed (Participants) | 177
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 174
  >=65 years | 3
Age Continuous [Mean (Standard Deviation); unit: years] | 51.9 (7.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111
  Male | 66
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 171
  More than one race | 4
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Summary of Treatment Emergent Adverse Events (TEAE).
Description: All adverse events reported were treatment emergent. Therefore, events that had a date of onset, or worsening, on or after the start of the open-label drug and up to 14 days after the last dose (for non-serious events) or up to 30 days after the last dose (for SAEs) were summarized. Any abnormal clinically significant changes in physical examination, medical history, clinical laboratory testing, 12-lead ECG, and standard EEG testing were captured as adverse events.
Time Frame: over 7 years (2004-2011)
Population: Safety Population. No imputation for missing data
Measure: Number; unit: participants
Groups:
- Fampridine-SR b.i.d.: All subjects (N=177) received 10mg b.i.d. Tablets.
  (N=175) subjects received 15mg b.i.d and (N=7) subjects received 20mg b.i.d at some point in the study.
Arm/Group | Fampridine-SR b.i.d.
Number analyzed (Participants) | 177
participants
  Patients with Any AE | 176 (99.4)
  Patients with Any Serious AE | 65 (36.7)
  Patients with Any Possibly/Probably Related AE | 102 (41.8)
  Patients withdrawn due to AE | 34 (15.3)
  Patients who Died | 5 (2.3)
  Maximum Severity/Patients with Any TEAE -Mild | 10 (8.5)
  Maximum Severity/Patients with Any TEAE -Moderate | 66 (38.4)
  Maximum Severity/Patients with Any TEAE -Severe | 100 (47.5)

2. Secondary Outcome: Timed 25 Foot Walk (T25FW)
Time Frame: Screening visit, visit 4, every 12 weeks thereafter, Last Regular Visit, Follow Up Visit and Early Termination Visit
Population: ITT Population. No imputation for missing data
Measure: Mean (Standard Deviation); unit: feet/second
Arm/Group | Fampridine-SR b.i.d.
Number analyzed (Participants) | 177
feet/second
  (N=153) Baseline | 1.87 (0.94)
  (N=1) >0-8 Weeks | 1.98 (NA) — 1 patient analyzed at time point therefore standard deviation not applicable
  (N=134) >8-16 Weeks | 2.09 (1.03)
  (N=141) >16-42 Weeks | 2.02 (1.04)
  (N=127) >42-68 Weeks | 1.82 (0.10)
  (N=111) >68-94 Weeks | 1.85 (1.05)
  (N=103) >94-120 Weeks | 1.77 (1.05)
  (N=92) >120-146 Weeks | 1.88 (0.10)
  (N=86) >146-172 Weeks | 1.84 (1.06)
  (N=76) >172-198 Weeks | 1.93 (1.34)
  (N=66) >198-224 Weeks | 1.82 (1.07)
  (N=56) >224-250 Weeks | 2.05 (1.16)
  (N=52) >250-276 Weeks | 2.03 (1.08)
  (N=54) >276-302 Weeks | 1.96 (1.09)
  (N=50) >302-328 Weeks | 1.98 (1.12)
  (N=10) >328-354 Weeks | 1.89 (1.57)

3. Secondary Outcome: Subject Global Impression (SGI)
Description: The patient was asked to complete a Subject Global Impression (SGI) questionnaire at Visit 1 and every study visit thereafter except the Follow-up visit. This questionnaire asked the patient to rate the effects of the investigational drug on his/her physical well-being during the preceding week, using a 1 to 7 point scale (1 = terrible, 7 = delighted)
Time Frame: visit 1 and every clinic visit
Population: ITT Population. No imputation for missing data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fampridine-SR b.i.d.
Number analyzed (Participants) | 177
units on a scale
  (N=176) >0-8 Weeks | 4.79 (0.89)
  (N=168) >8-16 Weeks | 4.70 (1.31)
  (N=163) >16-42 Weeks | 4.71 (1.09)
  (N=148) >42-68 Weeks | 4.42 (1.09)
  (N=137)>68-94 Weeks | 4.67 (1.11)
  (N=128) >94-120 Weeks | 4.70 (1.17)
  (N=124) >120-146 Weeks | 4.73 (1.21)
  (N=114) >146-172 Weeks | 4.76 (1.29)
  (N=102) >172-198 Weeks | 4.84 (1.27)
  (N=91) >198-224 Weeks | 5.15 (1.15)
  (N=88) >224-250 Weeks | 5.10 (1.29)
  (N=84) >250-276 Weeks | 5.04 (1.16)
  (N=81) >276-302 Weeks | 4.91 (1.47)
  (N=74) >302-328 Weeks | 5.28 (1.21)
  (N=12) >328-354 Weeks | 5.08 (1.40)

4. Secondary Outcome: Clinician Global Impression of Change (CGIC)
Description: The CGIC was based on the Investigator's overall impression of the patient's neurological status and general state of health related to his or her participation in the study, specifically in regard to signs and symptoms associated with MS. Neurological status was rated according to a 1 to 7 point scale (1 = very much improved, 7 = very much worse)
Time Frame: visit 1 and every clinic visit
Population: ITT Population. No imputation for missing data
Measure: Median (Standard Deviation); unit: units on a scale
Arm/Group | Fampridine-SR b.i.d.
Number analyzed (Participants) | 177
units on a scale
  (N=176) >0-8 Weeks | 3.37 (0.59)
  (N=168) >8-16 Weeks | 3.47 (0.97)
  (N=163) >16-42 Weeks | 3.60 (0.83)
  (N=148) >42-68 Weeks | 3.80 (0.89)
  (N=137) >68-94 Weeks | 3.83 (0.89)
  (N=128) >94-120 Weeks | 3.76 (0.89)
  (N=124) >120-146 Weeks | 3.70 (0.98)
  (N=116) >146-172 Weeks | 3.96 (1.05)
  (N=102) >172-198 Weeks | 3.89 (0.82)
  (N=92) >198-224 Weeks | 3.75 (1.02)
  (N=87) >224-250 Weeks | 3.79 (0.83)
  (N=83) >250-276 Weeks | 3.87 (1.11)
  (N=80) >276-302 Weeks | 4.29 (1.28)
  (N=73) >302-328 Weeks | 4.27 (1.34)
  (N=13) >328-354 Weeks | 3.81 (1.75)

5. Secondary Outcome: Expanded Disability Status Scale (EDSS)
Description: Based on the baseline neurological exam, each patient was scored according to the Expanded Disability Status Scale, which rates disability on a 0 to 10 scale (0 = normal neurologic examination, 10 = death)
  *EDSS assessments were not well synchronized to study period because of wide differences in interval between screening and initiation
Time Frame: Screening visit, visit 6 and every 24 months thereafter
Population: ITT Population. No imputation for data missing
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fampridine-SR b.i.d.
Number analyzed (Participants) | 177
units on a scale
  (N=166) Baseline | 6.04 (1.09)
  (N=92) >8-16 Weeks | 6.14 (0.91)
  (N=114) >42-68 Weeks | 6.26 (1.20)
  (N=56) >146-172 Weeks | 6.03 (1.31)

ADVERSE EVENTS:
Arm/Group | Fampridine-SR b.i.d. (Twice Daily)
Serious Adverse Events (participants affected / at risk) | 65/177
Other Adverse Events (participants affected / at risk) | 176/177
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fampridine-SR b.i.d. (Twice Daily) (N=177)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Angina Unstable (Cardiac disorders) | 1 (1)
Aortic Rupture (Vascular disorders) | 1 (1)
Appendicitis Perforated (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Back Injury (Injury, poisoning and procedural complications) | 1 (1)
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bowen's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Brain Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Bronchioloalveolar Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Calculus Bladder (Renal and urinary disorders) | 1 (1)
Cellulitis (Infections and infestations) | 3 (4)
Cervical Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest Pain (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Complex Partial Seizures (Nervous system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Convulsion (Nervous system disorders) | 2 (2)
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Depressed Level of Consciousness (Nervous system disorders) | 1 (1)
Device Malfunction (Injury, poisoning and procedural complications) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Drug Toxicity (Injury, poisoning and procedural complications) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3)
Femur Fracture (Injury, poisoning and procedural complications) | 2 (2)
Haemorrhage (Vascular disorders) | 1 (1)
Haemorrhage Intracranial (Nervous system disorders) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1)
Hepatic Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hip Fracture (Injury, poisoning and procedural complications) | 3 (3)
Hypertension (Vascular disorders) | 1 (1)
Influenza (Infections and infestations) | 2 (2)
Influenza Like Illness (General disorders) | 1 (1)
Kidney Infection (Infections and infestations) | 1 (1)
Limb Injury (Injury, poisoning and procedural complications) | 1 (1)
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Mania (Psychiatric disorders) | 1 (1)
Mental Status Changes (Psychiatric disorders) | 1 (1)
Multiple Sclerosis (Nervous system disorders) | 5 (5)
Multiple Sclerosis Relapse (Nervous system disorders) | 12 (15)
Muscle Spasticity (Nervous system disorders) | 3 (3)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Neurogenic Bowel (Gastrointestinal disorders) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 1 (1)
Oedema Peripheral (General disorders) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1)
Orthostatic Hypotension (Vascular disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Paraparesis (Nervous system disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Postoperative Wound Infection (Infections and infestations) | 1 (1)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostatic Abscess (Infections and infestations) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Pyrexia (General disorders) | 2 (2)
Rectocele (Gastrointestinal disorders) | 1 (1)
Renal Cell Carcinoma Stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1)
Renal Failure Acute (Renal and urinary disorders) | 1 (1)
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rib Fracture (Injury, poisoning and procedural complications) | 1 (1)
Sepsis (Infections and infestations) | 4 (4)
Sinusitis (Infections and infestations) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Throat Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tibia Fracture (Injury, poisoning and procedural complications) | 1 (1)
Trigeminal Neuralgia (Nervous system disorders) | 1 (1)
Urethral Injury (Injury, poisoning and procedural complications) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 7 (9)
Urosepsis (Infections and infestations) | 3 (4)
Uterine Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Visual Disturbance (Eye disorders) | 1 (1)
Wound Infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fampridine-SR b.i.d. (Twice Daily) (N=177)
Adverse Drug Reaction (General disorders) | 19 (26)
Anxiety (Psychiatric disorders) | 13 (13)
Arthralgia (Musculoskeletal and connective tissue disorders) | 34 (49)
Asthenia (General disorders) | 32 (44)
Back Pain (Musculoskeletal and connective tissue disorders) | 30 (48)
Balance Disorder (Nervous system disorders) | 17 (24)
Blood Cholesterol Increased (Investigations) | 13 (15)
Blood Creatine Phosphokinase Increased (Investigations) | 11 (14)
Blood Triglycerides Increased (Investigations) | 9 (9)
Bronchitis (Infections and infestations) | 10 (14)
Cataract (Eye disorders) | 10 (16)
Cellulitis (Infections and infestations) | 9 (12)
Constipation (Gastrointestinal disorders) | 22 (30)
Contusion (Injury, poisoning and procedural complications) | 20 (33)
Cystitis (Infections and infestations) | 9 (14)
Depression (Psychiatric disorders) | 28 (29)
Diarrhoea (Gastrointestinal disorders) | 18 (24)
Dizziness (Nervous system disorders) | 29 (40)
Dyspepsia (Gastrointestinal disorders) | 10 (14)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 (18)
Erythema (Skin and subcutaneous tissue disorders) | 9 (10)
Excoriation (Injury, poisoning and procedural complications) | 10 (13)
Fall (Injury, poisoning and procedural complications) | 75 (157)
Fatigue (General disorders) | 39 (53)
Fungal Infection (Infections and infestations) | 18 (20)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 10 (11)
Headache (Nervous system disorders) | 40 (58)
Hypertension (Vascular disorders) | 20 (21)
Hypoaesthesia (Nervous system disorders) | 15 (19)
Influenza (Infections and infestations) | 14 (17)
Insomnia (Psychiatric disorders) | 52 (64)
Joint Sprain (Injury, poisoning and procedural complications) | 10 (10)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 11 (15)
Micturition Urgency (Renal and urinary disorders) | 14 (14)
Mobility Decreased (Musculoskeletal and connective tissue disorders) | 26 (32)
Multiple Sclerosis (Nervous system disorders) | 20 (23)
Multiple Sclerosis Relapse (Nervous system disorders) | 43 (68)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 31 (40)
Muscle Spasticity (Nervous system disorders) | 41 (47)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 45 (79)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 16 (19)
Myalgia (Musculoskeletal and connective tissue disorders) | 13 (15)
Nasopharyngitis (Infections and infestations) | 23 (32)
Nausea (Gastrointestinal disorders) | 24 (25)
Neck Pain (Musculoskeletal and connective tissue disorders) | 10 (11)
Nervousness (Psychiatric disorders) | 9 (10)
Oedema Peripheral (General disorders) | 40 (52)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 10 (10)
Pain (General disorders) | 16 (19)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 24 (37)
Paraesthesia (Nervous system disorders) | 23 (31)
Procedural Pain (Injury, poisoning and procedural complications) | 11 (15)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (11)
Pyrexia (General disorders) | 14 (17)
Rash (Skin and subcutaneous tissue disorders) | 18 (21)
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 11 (12)
Sinusitis (Infections and infestations) | 12 (14)
Skin Laceration (Injury, poisoning and procedural complications) | 15 (18)
Tremor (Nervous system disorders) | 15 (17)
Upper Respiratory Tract Infection (Infections and infestations) | 33 (61)
Urinary Incontinence (Renal and urinary disorders) | 10 (10)
Urinary Retention (Renal and urinary disorders) | 9 (9)
Urinary Tract Infection (Infections and infestations) | 84 (280)
Vertigo (Ear and labyrinth disorders) | 10 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor (Acorda) has right to review and comment on proposed publications within a specified time frame, up to 60 days; multi-center trials require joint publication unless specifically permitted otherwise.